CLINICAL TRIAL: NCT03786120
Title: The Efficacy of Lower Dose Zolpidem for Achieving Satisfactory Sleep in Women With Disordered Sleep
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Vitae Industries, Inc (Unknown)
Responsible Party: Principal Investigator, Angela Jarman, Teaching Fellow, Rhode Island Hospital
Other Study IDs: Ambien Study
Record Dates: First submitted 2018-01-24; First posted 2018-12-24 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Zolpidem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: First 25 subjects
  Interventions: Drug: Zolpidem
- 2: Second cohort of 25 subjects
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Drug: Zolpidem — PO sleep aid in various doses

SUMMARY:
Sleep difficulties are very common in adults in the U.S. today. Zolpidem (Ambien) is often prescribed as a first line agent to treat sleep difficulties in patients presenting with sleep related complaints to Primary Care Practitioners (PCP's). Zolpidem is currently available in two doses, 10 and 5 mg. These doses were developed in clinical studies carried out primarily on men. The first dose made clinically available, 10 mg, resulted in morbidity and mortality in many women because women metabolize Zolpidem at a slower rate than men, thus the half-life is longer. Women taking Zolpidem often had morning drowsiness, persistent sleepiness, and difficulty with tasks requiring coordination and judgement, such as motor vehicle operation. There were a number of well publicized motor vehicle crashes and fatalities attributed to Zolpidem, mostly among women. The company then produced a 5 mg dose; however, some women still reported side effects at the lower dose, suggesting persistent drug levels in the morning, when the drug purportedly should have been cleared from the body. These women would likely benefit from a lower dose, a dose personalized for their individual metabolisms and sleep difficulties. Lower doses of Zolpidem are only available from compounding pharmacies, which are not common, are expensive, do not take many insurances, and are not offered as an option to most patients. Vitae Industries, Inc. is a start-up tech company located in Providence, founded by a Brown University graduate, a chemical engineer, who has developed technology that can provide precisely varied amounts of drug for specific and variable personalized patient dosing. Personalized medicine is an area of great research and clinical interest to the medical community at large and the Brown University Medical School in particular. Brown also has a growing focus on issues of sex and gender in the rendering of clinical medical care. This technology has the potential to address both of these areas, providing the possibility of very specific, tailored drug dosing for men and women. This research was developed as a proof of concept study which will be carried out as a collaboration between Brown University Medical School/Lifespan physicians and the technical staff at Vitae Industries, Inc.. This work will be foundational and will serve as the medical and scientific justification for Vitae Industry's providing patient specific dosing of medications. For the purposes of this study, the medication to be tested, Zolpidem (Ambien) will be compounded by a licensed compounding Rhode Island pharmacy, PhusionRx, using standardized approaches to compounding and formulating pharmaceutical products. This study will use low doses of Zolpidem formulated by the licensed compounding pharmacy, PhusionRx. The investigators will provide graduated doses of Zolpidem to women participants meeting inclusion criteria who present to their primary care physician complaining of difficulty achieving satisfactory sleep. Participants will start at a dose of 0.5 mg of Zolpidem. Each day the quality of their sleep will be assessed by self-report. If they have not achieved satisfactory sleep at the starting dose of 0.5 mg, the will increase their dose daily by 0.5 mg until they reach the standard 5 mg dose or satisfactory sleep is achieved.

ELIGIBILITY:
Inclusion Criteria:

* biologically female
* age 18-65
* English speaking
* difficulty sleeping

Exclusion Critieria:

* diagnosed significant cardiac, pulmonary, neuromuscular, hepatic, renal or major psychiatric disease (as ascertained by the study physicians)
* diagnosed sleep pathology such as sleep apnea or prior work-up for sleep pathology
* recent (two weeks prior) treatment of any kind for sleep disorder including herbal or over the counter treatments, psychiatric medications including anxiolytics except for SSRI's.
* pregnant or trying to become pregnant

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Health Women with Disordered Sleep
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 7 days
  This will be based on the sleep journal

SECONDARY OUTCOMES:
Side Effects | 7 days
  Including daytime drowsiness, night walking/eating

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Becker, MD, Principal Investigator — Lifespan
Locations (1):
- rhode island Hospital, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT03786120/ICF_000.pdf